CLINICAL TRIAL: NCT01978132
Title: Primary Hyperaldosteronism and Endothelial Ischemia-reperfusion Injury
Brief Title: Primary Hyperaldosteronism and Ischemia-reperfusion Injury
Acronym: PHA-FMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL45381.091.13
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-04

CONDITIONS: Primary Hyperaldosteronism
Keywords: primary hyperaldosteronism; primary hypertension; forearm ischemia-reperfusion; (reduction) in brachial artery FMD; endothelial ischemia-reperfusion injury
MeSH Terms: conditions — Hyperaldosteronism; Essential Hypertension | interventions — Reperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary hyperaldosteronism (Active Comparator): patients with primary hyperaldosteronism will be subjected to the intervention forearm ischemia and reperfusion (20 minutes of forearm ischemia and 20 minutes of reperfusion).
  Primary endpoint is the reduction in brachial FMD by forearm ischemia-reperfusion, as a measure of endothelial ischemia-reperfusion injury
  Interventions: Procedure: forearm ischemia and reperfusion
- Primary hypertension (Placebo Comparator): Patients with primary hypertension (PHA excluded)will be subjected to 20 minutes of forearm ischemia and 20 minutes of reperfusion.
  Primary endpoint is the reduction in brachial FMD by forearm ischemia-reperfusion, as a measure of endothelial ischemia-reperfusion injury
  Interventions: Procedure: forearm ischemia and reperfusion

INTERVENTIONS:
Procedure: forearm ischemia and reperfusion — both arms will be subjected to 20 minutes of forearm ischemia and 20 minutes of reperfusion.

SUMMARY:
Patients with primary hyperaldosteronism experience more cardiovascular events compared to patients with primary hypertension, independent of the blood pressure level.

In this research we hypothesize that patients with primary hyperaldosteronism are more susceptible to ischemia-reperfusion injury.

DETAILED DESCRIPTION:
Patients with PHA have an increased risk of cardiovascular events, independent of blood pressure level. Also in patients suffering a myocardial infarction, circulating aldosterone levels are associated with increased mortality. In animal models of myocardial infarction, the administration of exogenous aldosterone increased infarct size, although other studies did not report this effect. In similar models, antagonists of the mineralocorticoid receptor (MR) reduced infarct size, which was completely abolished in ecto-5'-nucleotidase (CD73, the enzyme that catalyses extracellular formation of the endogenous nucleoside adenosine) and adenosine receptor knock-out mice. Therefore, we hypothesize that patients with PHA have an increased susceptibility for ischemia-reperfusion (IR)-injury due to down-regulation of the enzyme CD73. We will use the reduction in brachial flow-mediated dilation (FMD) by forearm IR as a well-validated endpoint for (endothelial) IR-injury.

ELIGIBILITY:
Inclusion Criteria patients with primary hyperaldosteronism:

* Age 18-75 years
* Confirmed primary hyperaldosteronism (aldosterone >0.28 nmol/l after salt loading)
* Serum potassium ≥ 3.5 mmol/L (with or without potassium supplementation)
* Written informed consent

Inclusion Criteria patients with primary hypertension:

* Age 18-75 years
* Primary hypertension
* Baseline aldosterone <0.30 nmol/l and aldosterone-renin-ratio<0.09
* Serum potassium ≥ 3.5 mmol/L
* Written informed consent

Exclusion Criteria for both arms (patients with primary hyperaldosteronism and patients with primary hypertension:

* Smoking
* History of atherosclerotic disease (myocardial infarction (MI), stroke, or peripheral vascular disease)
* Not possible to change the antihypertensive medication into only diltiazem with or without hydralazine, according to the treating physician.
* Not possible to temporarily interrupt statin treatment, if the patient use statins, according to the treating physician.
* Severe renal dysfunction (MDRD < 30 ml/min)
* Second/third degree AV-block on electrocardiography
* Cardiac failure
* Diabetes Mellitus
* Use of acetylsalicylic acid and NSAID's theophylline, and dipyridamole

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
brachial FMD | 1 day morning
  primary outcome measure is the reduction in brachial artery FMD after 20 minutes of forearm ischemia and 20 minutes of reperfusion in patients with primary hyperaldosteronism (compared to patients with primary hypertension)

SECONDARY OUTCOMES:
CD73 and adenosine | one day morning (just before FMD experiment)
  Blood will be drawn to determine circulating adenosine concentration and the CD73 activity on mononuclear cells

OTHER OUTCOMES:
aldosterone and renin | 1 day
  Just before the FMD experiment, blood will be drawn for aldosterone and renin levels. These levels will not be determined, unless the brachial artery FMD after ischemia and reperfusion is significantly reduced in patients with primary hyperaldosteronism. We will store the plasma and serum at -20 C. If applicable, the aldosterone and aldosterone-to-renin ratio will be determined to correlate the primary outcome measure to the aldosterone and ARR levels.
leukocyte telomere length (LTL) | 1 day
  We will measure LTL in 12 patients with PHA and 12 patients with EHT to assess wether aldosterone excess increases telomere shortening in patients with PHA

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands